CLINICAL TRIAL: NCT07226375
Title: Comparison of Endoscopic Tissue Cutting and Abdominal Extraction Device With Conventional Cold Scalpel
Brief Title: Endoscopic Tissue Cutting and Abdominal Extraction Device vs. Conventional Cold Scalpel
Acronym: SOLENDO-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBAP.2023.003
Record Dates: First submitted 2024-10-25; First posted 2025-11-10 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Hysterectomy
Keywords: laparoscopic hysterectomy; morcellation; tissue extraction
MeSH Terms: interventions — Device Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Endoscopic Tissue Cutting and Abdominal Extraction Device (Experimental): In the cases included in the group, vaginal morcellation will be performed with an endoscopic tissue cutting and removal device after laparoscopic hysterectomy.
  Interventions: Device: Vaginal tissue morcellation with extraction device
- Conventional Cold Scalpel (Active Comparator): In the cases included in the group, vaginal morcellation will be performed with a cold scalpel after laparoscopic hysterectomy.
  Interventions: Device: Vaginal tissue morcellation with scalpel

INTERVENTIONS:
Device: Vaginal tissue morcellation with extraction device — Vaginal tissue morcellation after laparoscopic hysterectomy with Endoscopic Tissue Cutting and Abdominal Extraction Device
  Arms: Endoscopic Tissue Cutting and Abdominal Extraction Device
Device: Vaginal tissue morcellation with scalpel — Vaginal tissue morcellation after laparoscopic hysterectomy with cold scalpel
  Arms: Conventional Cold Scalpel

SUMMARY:
The aim of the study is to compare the surgical tissue removal success of the endoscopic tissue cutting device, which was designed by the conductor and developed with the support of TUBITAK-1512 project and for which Turkish and European patent applications were made, with the conventional cold scalpel. Laparoscopic surgeries are performed through incisions ranging from 0.5 cm to 1 cm. After the operation, much larger masses need to be removed from the abdomen compared to these incisions. Currently, in laparoscopic surgery, masses are removed from the abdomen by cutting them into pieces with a scalpel, using electrical devices called power morcellators that are used to cut the tissue/mass with rotational movement and remove it from the abdomen, and directly removing the mass from the abdomen through an incision made as large as the size of the mass. Trying to remove large tissues/mass by dissecting them with a scalpel through incisions that are 1.5-2 cm wide and limit the surgeon's range of motion is quite laborious, tiring, time-consuming and risky. In the use of Power Morcellator disintegrator devices, there is a risk of the pieces of the mass spreading into the abdomen while cutting and separating the tissue/mass that is being removed into small pieces due to the rotational movement in the working principle. In operations where the Power Morcellator device is used, if the removed tissue is malignant (cancerous), the patient faces the risk of metastasis spreading to the entire abdomen. Due to these risks, the use of power morcellator devices has been completely banned in the United States, and in European Union countries, it has been required that the device be operated in protective bags. The invention is a medical device that will allow large masses to be removed quickly, safely and easily through small incisions in closed surgeries. The device offers an effective solution to the problems of the current technique.

Within the scope of the study, the morcellator scissors and the scalpel, which are designed and started to be mass-produced, will be compared in the morcellation (removal by separating into pieces) process to be performed during the removal of the mass from the vagina after laparoscopic hysterectomy surgeries, and the morcellation time, possible complications and the possible effects of the device to be used on the case will be investigated.

DETAILED DESCRIPTION:
Laparoscopic surgeries are performed through incisions ranging from 0.5 cm to 1 cm in width. After the operation, masses that are much larger than these incisions need to be removed from the abdomen. The process of removing masses from the abdomen is a difficult and time-consuming process, often taking longer than the operation itself and forcing surgeons to perform open surgery. Therefore, patients are deprived of the comfort of closed surgery and experience disadvantages such as risk of infection, pain, and staying away from work and social life for a long time. The invention allows tissues/mass that are intended to be removed from the abdomen in laparoscopic surgery and are larger in size than the incisions where the operation is performed to be removed from the abdomen through these incisions. The designed device offers a fast, easy and reliable alternative to removing tissues or masses from the abdomen, which is the most time-consuming and tiring stage of laparoscopic surgery.

Currently, removing masses from the abdomen in laparoscopic surgery;

* Cutting into pieces with a scalpel,
* Using electrical devices called morcellators that are used to cut the tissue/mass with a rotational movement and take it out of the abdomen,
* It is done by directly removing the mass from the abdomen through an incision made as large as the size of the mass.

Trying to break up large tissues/mass with a scalpel through 1.5-2 cm wide holes/incisions that limit the surgeon's field of movement is quite laborious, tiring, time-consuming and risky in terms of patient health. This process can extend the duration of the surgery by 60 to 90 minutes (Nieboer et al., 2009). In addition, the risk of injury or damage to surrounding tissues is high due to the aforementioned procedures.

In the use of morcellator disintegrating devices, there is a risk that the tissue/mass that is being removed will spread/scatter into the abdomen in small pieces due to the rotational movement in the operating principle. In operations where the morcellator device is used, if the removed tissue is malignant (cancerous), the patient is at risk of metastasis spreading to the entire abdomen. Due to the bitter experiences, the use of this device has been banned in the United States and in European Union countries, it has been required to be used in sterile bags. However, even the use of these bags cannot completely prevent the spread of tissue into the abdomen.

Another way to remove the mass from the abdomen at the end of the operation is to make a large incision in the abdomen. This incision eliminates all the advantages of laparoscopic surgery, increases the patient's pain and prolongs the hospital stay, increases the cost of the operation, creates an infection risk and therefore delays the patient's return to work/social life.

With the invention and project, the mass to be removed from the abdomen after the laparoscopic operation can be removed without an additional abdominal incision in the hysterectomy (uterus removal) surgery; In myomectomy or adnexal mass surgeries, it will be shown that it can be easily removed by cutting into pieces through a 3 cm incision made at the top of the vagina. With the designed device, the tissue/mass can be quickly and safely removed from the abdomen with repetitive movements. Since large-sized tissues/mass can be removed from the abdomen through a maximum 3 cm incision with the advantage provided by the invention, patients are protected from the possible risks of a large incision. Since the invention cuts the tissue/mass directly (does not make a rotation movement like the morcellator device) and is designed to keep the cut piece in its own chamber, there is no risk of the tissue/mass spreading into the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Planned laparoscopic hysterectomy
* Estimated uterine weight of 500 g or more

Exclusion Criteria:

* Sexual inactivity

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 84 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Morcellation Time | From placement of uterus in retrieval bag to complete removal of specimen, measured in minutes (approximately 0-30 minutes).
  The time required for complete vaginal morcellation of the uterus, measured from the placement of the uterus into the retrieval bag until complete specimen removal. A shorter duration indicates higher procedural efficiency.

SECONDARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) Score | Baseline (within 1 week before surgery) and 6 months after operation.
  The change in total Female Sexual Function Index (FSFI) score between the preoperative and postoperative periods will be assessed to evaluate the impact of vaginal morcellation technique on sexual function.
  The FSFI is a validated questionnaire assessing sexual function in six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain.
  Total scores range from 2 to 36, with higher scores indicating better sexual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared at this stage to protect intellectual property rights related to the patented device. Deidentified data may be made available upon reasonable request after study completion